CLINICAL TRIAL: NCT00554294
Title: Promoting Water Consumption for Prevention of Overweight in School Children in a Controlled Intervention Trial
Acronym: trinkfit
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Research Institute of Child Nutrition, Dortmund (Other)
Responsible Party: Research Institute of Child Nutrition, Dortmund, Research Institute of Child Nutrition, Dortmund
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 05HS026
Record Dates: First submitted 2007-11-05; First posted 2007-11-06 (Estimated); Results first posted 2009-07-16 (Estimated); Last update posted 2009-07-16 (Estimated); Status verified 2009-05

CONDITIONS: Overweight
Keywords: children; primary prevention; environmental change; behavioural change; school setting; changing of drinking habits; promotion of drinking tap water
MeSH Terms: conditions — Overweight | interventions — Environment

ARMS (2):
- Control group (No Intervention): Control schools had school curriculum as usual and did not receive environmental intervention.
- Intervention group (Experimental): Intervention schools received water dispensers, drinking bottles and lessons as intervention.
  Interventions: Behavioral: environmental and behavioral change

INTERVENTIONS:
Behavioral: environmental and behavioral change — In intervention schools a water dispenser was installed and children received water bottles as environmental intervention. Children also received a 6-hour-curriculum about the importance of water for the body that were held by the teachers.
  Arms: Intervention group

SUMMARY:
A major goal in public health is to find effective, feasible and simple programs for overweight prevention among children. This controlled intervention study evaluates a simple environmental and behavioral modification for its efficacy in preventing overweight of children in the school setting. The intervention strategy focuses solely on the promotion of drinking tap water. The study was conducted in 32 elementary schools including about 3000 children in two German cities over 1 school year.

DETAILED DESCRIPTION:
Soft drinks and other caloric beverages are supposed to be involved in the development of overweight and obesity in children. The intervention strategy of our study was to promote water consumption by facilitating access to tap water in schools assuming a concomitant decrease in caloric soft drinks at least at school. The environmental modification of installing a water dispenser at school and delivering a special bottle to each child in the intervention schools was supported by a few educational lessons. These lessons were held by the class teachers who received a prepared 6-hour curriculum dealing with the importance of water for the body and of water intake. For the study 17 randomly selected schools were assigned to the intervention group, 15 schools to the control group that did not receive any intervention. Body weight and height to calculate BMI as primary outcome were assessed at baseline and after the intervention period of 1 school year. As secondary outcome drinking and physical activity habits were evaluated at baseline and after the intervention. The water flow of the dispenser was measured at regular intervals. In addition, data of process evaluation was collected to measure acceptance and feasibility of the intervention in the school setting.

To analyze the efficacy of this primarily environmental and behavioral intervention, incidence and prevalence was compared between intervention and control group.

ELIGIBILITY:
Inclusion Criteria:

* All children in 2nd and 3rd grade of selected elementary schools

Exclusion Criteria:

* parental consent

Ages: 7 Years to 9 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 2950 (Actual)
Dates: Start 2006-04; Primary Completion 2007-06 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mathilde Kersting, PhD, Principal Investigator — Research Insitute of Child Nutrition

REFERENCES:
- [Result] Muckelbauer R, Libuda L, Clausen K, Toschke AM, Reinehr T, Kersting M. Promotion and provision of drinking water in schools for overweight prevention: randomized, controlled cluster trial. Pediatrics. 2009 Apr;123(4):e661-7. doi: 10.1542/peds.2008-2186. PMID 19336356
- [Derived] Muckelbauer R, Libuda L, Clausen K, Toschke AM, Reinehr T, Kersting M. Immigrational background affects the effectiveness of a school-based overweight prevention program promoting water consumption. Obesity (Silver Spring). 2010 Mar;18(3):528-34. doi: 10.1038/oby.2009.270. Epub 2009 Aug 27. PMID 19713953

RESULTS

PARTICIPANT FLOW:
Recruitment Details: second and third graders of participating schools
Groups:
- Control Group: Schools did not receive any intervention.
- Intervention Group: Schools received water fountains, drinking bottles and lessons as intervention.
Period: Overall Study
Arm/Group | Control Group | Intervention Group
Started | 1469 | 1721
Completed | 1309 | 1641
Not Completed | 160 | 80

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control Group | Intervention Group | Total
Number analyzed (Participants) | 1469 | 1721 | 3190
Age Continuous [Mean (Standard Deviation); unit: years] | 8.3 (0.7) | 8.3 (0.7) | 8.3 (0.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 734 | 853 | 1587
  Male | 735 | 868 | 1603
Prevalence of overweight [Number; unit: participants] — Overweight was defined according to the standard of the International Obesity Task Force
  participants
    overweight | 378 | 404 | 782
    non-overweight | 1091 | 1317 | 2408

OUTCOME MEASURES:

1. Primary Outcome: Overweight
Description: Prevalence of overweight defined acording to the criteria of the International Obesity Task Force (IOTF)
Time Frame: one school year
Measure: Number; unit: participants
Arm/Group | Control Group | Intervention Group
Number analyzed (Participants) | 1309 | 1641
participants | 683 | 385
Statistical Analysis 1: Comparison: Control Group vs Intervention Group; adjusted for overweight at baseline, age at baseline,sex and clustering by school; Test type: Superiority or Other; p < 0.05, Regression, Logistic; The Odds Ratio (OR) describes the probability ob beeing overweight of the intervention group compared to the control group (reference, denominator); Odds Ratio (OR) = 0.69, 95% CI [0.48 to 0.98]

2. Secondary Outcome: Intake of Drinks
Time Frame: one school year
Reporting Status: Not Posted

3. Secondary Outcome: Physical Activity and Inactivity
Time Frame: one school year
Reporting Status: Not Posted

4. Secondary Outcome: Water Flow of the Water Dispensers
Time Frame: one school year
Reporting Status: Not Posted

5. Secondary Outcome: Parameters of Process Evaluation (Acceptance, Feasibility)
Time Frame: 1,5 years
Reporting Status: Not Posted

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No